CLINICAL TRIAL: NCT04727658
Title: Linac FRACtionated Radiosurgical THALamotomy in Tremors : a Phase II Study
Brief Title: Linac FRACtionated Radiosurgical THALamotomie in Tremors (FRACTHAL)
Acronym: FRACTHAL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01
Record Dates: First submitted 2021-01-11; First posted 2021-01-27 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Essential Tremor; Parkinsonian Disorders
MeSH Terms: conditions — Essential Tremor; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: The study will be carried out according to a design by Simon in two stages (Simon, 1989).
  First step: 14 patients will be included in the study. When the 14th patient has been treated, the inclusions will be suspended for 1 year until analysis of the primary endpoint.
  • Second stage: 34 additional patients will be recruited for a total of 48 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiosurgical thalamotomy on GammaKnife (Experimental)
  Interventions: Radiation: Radiosurgical thalamotomy on GammaKnife

INTERVENTIONS:
Radiation: Radiosurgical thalamotomy on GammaKnife — fractional radiosurgical thalamotomy on an accelerator (3 sessions of 50 Gy at the isocenter )

SUMMARY:
Radiosurgical thalamotomy on GammaKnife has been shown to be effective in the management of tremors. However, several teams describe a significant risk of severe neurological complications. In addition, fitting the invasive frame and the need to travel to GammKnife centers often limit access to treatment in this population of elderly patients.

Linear accelerators have greatly improved their precision, now reaching that of GammaKnife. A possible alternative is therefore to treat patients on linear accelerators, without an invasive frame.

The objective of the FRACTHAL study is to assess the feasibility and safety of treatment of essential and / or parkinsonian tremor by fractional radiosurgical thalamotomy on a linear accelerator.

The main hypothesis of the FRACTHAL study is based on the fact that dividing the dose into 3 sessions will both protect healthy tissue around the target while maintaining therapeutic efficacy on the treatment target.

ELIGIBILITY:
Inclusion Criteria:

* patient with disabling essential tremor, dystonic and / or parkinsonian in one or more limbs superiors ;
* patient contraindicated or refusing deep brain stimulation ;
* patient ≥ 18 years old,
* women of childbearing potential must take effective contraception ;
* signature of informed consent ; p- atients who benefited from contralateral thalami c stimulation can be included in the study

Exclusion Criteria:

* brain irradiation history ;
* contraindication or inability to perform injected MRI ;
* life expectancy <12 months ;
* claustrophobic patient who cannot stand the radiotherapy mask ;
* abnormal anatomy of the thalamic region ;
* treatment with a trial drug within 30 days of entering the study ;
* presence of medical, psychological, social or geographic factors likely to modify the patient's compliance with the protocol under study or the monitoring or signing of the consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Treatment toxicity | 12 months
  The treatment will be considered toxic in the event of the appearance, within 12 months after treatment, of non-regressive toxicity of grade> 1 according to the NCI-CTCAE V5.0 scale (symptomatic neurological deficit interfering with daily activities), and that this deficit is related to the treatment.

SECONDARY OUTCOMES:
Treatment accuracy | At 6 and 12 months
  Measurement of the shift between the position of the treatment isocenter and the position of the hypersignal center visible on the injected MRI
Tremor improvement | At 3, 6 and 12 months
  It will be measured by decrease in FTM scale score for contralateral upper limb

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No
no data sharing is planned